CLINICAL TRIAL: NCT05220930
Title: The Effect of a Foot Bath Before Capillary Heel Blood Sampling on Pain and Procedure Time in Neonates: A Randomized Clinical Trial
Brief Title: Foot Bath for Heel Warming Before Heel Lance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta University of Applied Sciences (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IspartaUASNursingCare
Record Dates: First submitted 2022-01-12; First posted 2022-02-02 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-01

CONDITIONS: Nursing Caries
Keywords: Foot bath; Heel warming; Heel Lance; Newborn; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot bath for heel warming group (Experimental): In this study, in line with the literature, the attempt to apply heat with a foot bath will be carried out by immersing both legs of the newborn in a basin filled with 15-20 cm of water at 38-40C, 5 minutes before the heel blood collection, starting just below the knee level. The intervention will be applied while the newborn is held in an upright position on his mother's lap. Before piercing the heel, the heel will be wiped with a blanket and dried. After the intervention, blood collection from the heel will be performed by following the standard procedure steps that are routinely applied in the service.
  Interventions: Other: Foot bath for heel warming
- Ineffective heel warming with thermofor group (Other): Ineffective heel warming will be applied to the newborns in the control group with a thermofor containing 28C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service.
  Interventions: Other: Ineffective heel warming with thermofor

INTERVENTIONS:
Other: Foot bath for heel warming — In this study, in line with the literature, the attempt to apply heat with a foot bath will be carried out by immersing both legs of the newborn in a basin filled with 15-20 cm of water at 38-40C, 5 minutes before the heel blood collection, starting just below the knee level. The intervention will be applied while the newborn is held in an upright position on his mother's lap.
  Arms: Foot bath for heel warming group
Other: Ineffective heel warming with thermofor — Ineffective heel warming will be applied to the newborns in the control group with a thermofor containing 28C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service.
  Arms: Ineffective heel warming with thermofor group

SUMMARY:
Foot bath is a simple warm application method that creates a feeling of comfort and positive effects on health have been reported in the literature. There are studies reporting the benefits of footbath for different groups. However, no study has been found in the literature investigating the effect of foot bath for heel warming before heel stick procedure on pain, and procedure time. Foot bath to be applied during heel blood collection is a cost-effective and easy-to-apply method. This study aims to determine the effect of foot bath for heel warming before heel stick procedure on pain, and procedure time in healthy term newborns.

DETAILED DESCRIPTION:
Aim: This study aimed to determine the effect of foot baths applied before capillary heel blood sampling for newborn on pain level and procedure duration in term newborns.

Method: This study was planned as a randomized controlled, experimental, single-center study. The universe of the research will be term newborns whose heel blood samples will be taken within the scope of the Newborn Screening Program (NSP) in the Isparta Şehir Hospital Gynecology and Obstetrics III Service.

The sample size of the study was calculated based on the first hypothesis of the study with the G*Power 3.1 program. The sample of the study was determined as 80 healthy term newborn (40 control, 40 intervention).

Intervention: In this study, ineffective heel warming with thermofor will be applied to the control group and foot bath for heel warming will be applied to the intervention group.

Data collection instruments: Newborn Information Form (NIF), and NIPS (Neonatal Infant Pain Scale) will be used to collect data.

Data collection: In this study, the effectiveness of the intervention was pre-intervention/pre-evaluation (T1); It will be evaluated at four measurement points during the procedure (T2); 1 minute after the procedure (T3); and 5 minutes after the procedure (T4). Measurement points were determined in accordance with the literatüre. Heel blood collection will be video-recorded from the pre-evaluation stage (one minute before the intervention) until the 5th minute after the procedure. The video recording will be monitored by two independent evaluators who do not know the purpose of the study, and the NIPS scores at the measurement points and the processing time will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Born between 38-42 gestational weeks (term newborns)
* Newborns with a birth weight of 2500-4400 grams
* Newborns with stable physiological parameters and general condition
* Newborns with vitamin K and hepatitis B vaccine in the delivery room
* Newborns with eight or more Apgar scores in the first and fifth minutes

Exclusion Criteria:

* Newborns with problems during pregnancy, labor and postpartum
* Newborns with congenital anomaly
* Newborns receiving pharmacological or non-pharmacological pain management intervention before the procedure
* Newborns with receiving oxygen therapy
* Newborns with having undergone a surgical procedure
* Newborns with sepsis or suspected sepsis
* Newborns whose parents state that they want to leave the study while the study continues

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Prosedüre time measure | During the procedure
  The video recording will be monitored by two independent evaluators who do not know the purpose of the study, and the processing time will be recorded.

SECONDARY OUTCOMES:
NIPS (Neonatal Infant Pain Scale) | Pre-intervention/pre-evaluation (T1); during the procedure (T2); 1 minute after the procedure (T3); and 5 minutes after the procedure (T4).
  The NIPS (Neonatal Infant Pain Scale) was developed by Lawrence et al. in 1993 and tr into translated into Turkish by Akdovan in 1999 to assess pain. This scale consists of five behavioral indicators including facial expression, leg, movement, arm movement, crying and wakefulness, and one physiological indicator of respiratory rhythm. Total scores range from 0 to Higher scores show that the intensity of pain is higher. The internal consistency of NIPS was reported to be 0.95 before the transaction, 0.87 during the transaction, and 0.88 after the transaction. According to a study conducted by Akdovan et al. in 1999, the internal consistency coefficient of this scale using Cronbach's alpha was found to be between 0.83 and 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Fahriye PAZARCIKCI, PhD, Study Director — Isparta University of Applied Sciences; Ayla KAYA, PhD, Study Chair — Akdeniz University
Locations (1):
- Isparta University of Applied Sciences, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
N/O

REFERENCES:
- [Result] Shu SH, Lee YL, Hayter M, Wang RH. Efficacy of swaddling and heel warming on pain response to heel stick in neonates: a randomised control trial. J Clin Nurs. 2014 Nov;23(21-22):3107-14. doi: 10.1111/jocn.12549. Epub 2014 Jan 30. PMID 24476226
- [Result] Unal C, Welcome MO, Salako M, Abdullahi F, Abubakar NM, Pereverzev VA, Hartiningsih SS, Dane S. The effect of foot reflexotherapy on the dynamics of cortical oscillatory waves in healthy humans: An EEG study. Complement Ther Med. 2018 Jun;38:42-47. doi: 10.1016/j.ctim.2018.03.006. Epub 2018 Mar 20. PMID 29857878